

# Statistical Analysis Plan Part A, Part B, Part C and Part D Analysis

# A SINGLE/MULTIPLE ASCENDING DOSE PHASE 1 STUDY OF THE SAFETY, TOLERABILITY, AND PHARMACOLOGIC ACTIVITY OF BT200 IN NORMAL HUMAN VOLUNTEERS

Protocol: BT200-01 NCT #04103034

Confidential

Sponsor: Band Therapeutics, LLC



# **Table of Contents**

| 1. | OVER | VIEW | 6 |
|---|---|---|---|
| | 1.1<br>1.1.1<br>1.1.2<br>1.1.3 | Study Objectives Primary Objective Secondary Objective Exploratory Objectives | 6<br>6<br>6<br>6 |
| | 1.2 | Study Design | 6 |
| | 1.3<br>1.3.1<br>1.3.2<br>1.3.3 | Endpoints Primary Endpoint Secondary Endpoints Exploratory Endpoints | 7<br>7<br>8<br>8 |
| | 1.4 | Sample Size Calculation | 8 |
| | 1.5 | Flowchart and Schedules of Assessments | 8 |
| 2. | GENE | RAL CONSIDERATIONS | 18 |
| | 2.1 | Rationale | 18 |
| | 2.2 | Conduct of Analysis | 18 |
| | 2.3 | Statistical Software and Quality Control | 18 |
| | 2.4 | Applicable Standard Operating Procedures | 18 |
| | 2.5 | Blinding and Randomization | 19 |
| | 2.6 | Descriptive Analyses | 19 |
| | 2.7 | Inferential Analyses | 19 |
| | 2.8 | Center and Country Effect | 19 |
| | 2.9 | Handling Missing Data | 19 |
| | 2.10 | Protocol Deviations | 20 |
| | 2.11 | Medical Coding | 20 |
| | 2.12<br>2.12.1<br>2.12.2 | | 20<br>20<br>20 |
| | 2.13 | Subject Data Listings | 21 |
| | 2.14 | Columns in Tables | 21 |
| | 2.15 | Changes in the Conduct of the Study or Planned Analysis | 21 |
| | 2.16 | Effect of Covid-19 | 21 |
| 3. | OVER | ALL STUDY INFORMATION | 21 |
| 4. | BASE | LINE EVALUATION | 22 |
| | 4.1 | Data Points | 22 |
| | 4.2 | Derivations and Definitions | 22 |
| 5. | PHAR | MACOKINETICS / PHARMACODYNAMICS / BIOMARKER / IMMUNOGENICITY | 23 |



| | 5.1 | Pharmacokinetics | 23 |
|---|---|---|---|
| | 5.2 | Pharmacodynamics | 23 |
| | 5.3 | Biomarker | 23 |
| | 5.4 | Immunogenicity | 24 |
| 6. | SAFE | TY ANALYSIS | 24 |
| | 6.1 | Extent of Exposure | 24 |
| | 6.2<br>6.2.1<br>6.2.2 | Adverse Events and Bleeding Events<br>Data Points<br>Definitions and Derivations | 24<br>24<br>25 |
| | 6.3 | Laboratory Parameters | 26 |
| | 6.4 | Other Safety Parameters | 27 |
| 7. | LIST | OF TABLES, DATA LISTINGS AND FIGURES | 28 |
| | 7.1 | List of Tables | 29 |
| | 7.2 | List of Data Listings | 34 |
| | 7.3 | List of Figures | 37 |
| 8. | SHEL | LS OF TABLES, DATA LISTINGS AND FIGURES | 38 |



| | | Document | |
|---|---|---|---|
| Study | BT200-01 | | |
| Document | Statistical Analysis Plan | (SAP) | |
| Version | FINAL 3.0 | | |
| Date | 17-Sep-2020 | | |
| | Rev | ision History | |
| Version | Date | Reaso | on for Revision |
| FINAL 1.0 | 27-May-2020 | First version; | |
| FINAL 2.0 | 05-Jun-2020 | Patient overview and der added into the Topline Ar | mographic information tables nalyses |
| FINAL 3.0 | 17-Sep-2020 | events added, update of tables), additional bioma | 2 described, Topline Analyses |
| V V V V V | A | Approval | |
| Name | Role | Date | Signature |
| | | Author | |
| Lisa Hegele | Biostatistician | 17 Sep-2000 | linty |
| | As | ssign DMB | |
| Julian Larcher-Senn | Senior Biostatistician | 77- Sep - 2020 | Hoh |
| | Band Th | erapeutics, LLC | , |
| Jim Gilbert | Chief Executive Officer | 17 Sep2020 | or Colo |

Any photocopies taken of this document are not authorized or version controlled.



# **List of Abbreviations**

| ADA | Anti-drug antibody |
|------------------|--------------------------------------------------|
| AE | Adverse Event |
| AGES | Austrian Agency for Health and Food Safety GmbH |
| aPTT | Activated partial thromboplastin time |
| BA | Bioavailability |
| BDRM | Blind Data Review Meeting |
| BMI | Body Mass Index |
| CAT | Calibrated Automated Thrombogram |
| CI | Confidence Interval |
| CSP | Clinical Study Protocol |
| CSR | Clinical Study Report |
| DSMB | Data and Safety Monitoring Board |
| EC | Ethics Committee |
| ELISA | Enzyme-linked immunosorbent assay |
| FIH | First-In-Human |
| GP1b | Glycoprotein lb |
| IV | Intravenous |
| MAD | Multiple ascending dose |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NHV | Normal healthy volunteer |
| PD | Pharmacodynamic(s) |
| PFA | Platelet Function Analyzer |
| PK | Pharmacokinetic(s) |
| PP | Per-Protocol Per-Protocol |
| SAD | Single ascending dose |
| SC | Subcutaneous |
| SD | Standard deviation |
| SMQ | Standardized MedDRA Query |
| TLF | Tables, Listings and Figures |
| T <sub>max</sub> | Time to Maximum Plasma Concentration |
| VWF | Von Willebrand Factor |
| VWF:RiCo | Von Willebrand Factor:ristocetin co-factor assay |
| WHO | World Health Organization |



#### OVERVIEW

#### 1.1 Study Objectives

#### 1.1.1 Primary Objective

The primary objective of this study is to assess the clinical safety and tolerability of BT200 in normal human volunteers (NHVs).

#### 1.1.2 Secondary Objective

The secondary objectives of this study are to assess the human pharmacokinetics (PK) of BT200.

#### 1.1.3 Exploratory Objectives

The exploratory objectives of this study are to evaluate the human immunogenicity and Pharmacodynamics (PD) of BT200, as follows:

- To evaluate the presence of anti-drug antibodies (ADAs) against BT200
- To evaluate the human PD of BT200 with respect to von Willebrand Factor (VWF)-mediated platelet function
- To evaluate the human PK/PD relationship of BT200
- · To evaluate potentially useful biomarkers for future clinical trials
- To investigate the mechanism of action of BT200 on the human coagulation system

#### 1.2 Study Design

Study BT200-01 is a prospective, double-blind, randomized, placebo-controlled First-In-Human (FIH) study of BT200 in male and female NHVs with 4 sub-parts: Part A, a single ascending dose (SAD) study; Part B, a multiple ascending dose (MAD) study; Part C, a desmopressin challenge study; and Part D, a relative Bioavailability (BA) study.

Part A, the SAD study in NHVs, will be conducted according to an ascending dose cohort paradigm in which a unique cohort of NHVs will be treated at each single dose level. There will be 10 cohorts of NHVs (6:2 ratio of BT200:placebo; except for the sentinel pair [1:1 ratio]). Cohorts 1 through 10 will consist of 8 NHVs each, comprising 6 NHVs administered BT200 subcutaneous (SC) (0.18, 0.6, 1.8, 6.0, 12.0, 18.0, 24.0 by rapid SC injection, and 24.0, 36.0 mg, 48.0 mg by gradual SC infusion, respectively, for each cohort) and 2 NHVs administered placebo SC. Not all NHVs in a given cohort in Part A will be dosed on the same day: a sentinel pair (1 BT200, 1 placebo) will be dosed on the first day, then with a lag of at least 48 hours staggered groups roughly of 2 to 3 NHVs per day will be dosed thereafter. Cohorts 8-10 of Part A will be initiated only after submission and authorization of a Substantial Amendment to Ethics Committee (EC) and Austrian Agency for Health and Food Safety (AGES) summarizing the results of Cohorts 1-7.

Part B, the MAD study in NHVs, will also be conducted according to an ascending dose cohort paradigm. Part B will be initiated only after Substantial Amendment to EC and AGES has been submitted and authorized following completion of cohorts 8-10 of Part A and Part D. There will be 2 cohorts of NHVs, each consisting of 8 NHVs (6:2



ratio of BT200:placebo) in this part of the study. These cohorts will be administered an initial loading dose regimen of BT200 or placebo consisting of both a 2-hour IV infusion and an SC injection on Day 0, followed by 4 weekly (every 7 days) doses of BT200 or placebo by SC injection The dose levels in Part B are: a loading dose of 12.0 mg IV infused over 2 hours plus 12.0 mg SC injection followed by 4 maintenance doses of 12.0 mg SC injection in Cohort 13; a loading dose of 24.0 mg IV infused over 2 hours plus 24.0 mg SC injection followed by 4 maintenance doses of 24.0 mg SC injection in Cohort 14. Not all subjects in each of the cohorts of Part B will be dosed on the same day; rather, they will be dosed in staggered groups roughly of 2 to 3 subjects per day.

Part C, the desmopressin challenge will be initiated only after a Substantial Amendment to EC and AGES has been submitted and authorized following cohorts 8-10 of Part A and Part D. Part C will consist of a single cohort, Cohort 12, of 8 NHVs (6:2 ratio of BT200:placebo, plus desmopressin challenge) in this part of the study. Six subjects in Cohort 12 will be administered a single dose of 48.0 mg BT200 SC injection and 2 subjects administered a single dose of placebo on Day -4 as an SC injection All subjects will then be administered an intravenous (IV) infusion of 0.3  $\mu$ g/kg desmopressin over 30 minutes on Day 0 approximately 96 hours after the single dose of BT200 or placebo SC (i.e., at the predicted time to maximum plasma concentration [T<sub>max</sub>] for BT200).

Part D, the relative BA crossover, will be initiated only after a Substantial Amendment to EC and AGES has been submitted and authorized following cohorts 1-7 of Part A. Part D will consist of 1 cohort of NHVs, consisting of 8 NHVs (6:2 ratio of BT200:placebo) administered a single IV dose of BT200 of 24.0 and 2 NHVs administered a single dose of placebo IV over 24 hours on Day 0.. Part D could include NHVs who have previously participated in Part A.

Firstly Part A (cohorts 1-7), secondly Part A (cohorts 8-10) and Part D, and finally Part C and Part B will be conducted sequentially. There will be a DSMB safety review after dosing of NHVs in Cohorts 1-7 of Part A is completed before Cohorts 8-10 of Part A are initiated; again after Cohorts 8-10 of Part A and Part D before Part C and Part B is initiated. The safety data provided to the DSMB and the resulting DSMB opinion will be submitted as a Substantial Amendment to EC and AGES prior to initiating Cohorts 8-10 of Part A and Part D; again prior to initiating Part C and Part B.

#### 1.3 Endpoints

#### 1.3.1 Primary Endpoint

Overall safety and tolerability of BT200, assessed in terms of:

- Serious, drug-related adverse events (AEs)
- Premature terminations due to drug-related AEs
- Patterns of serious or non-serious, drug-related AEs, and/or clinically relevant laboratory abnormalities,
   vital signs, ECGs, or physical findings suggestive of one or more specific target organs for toxicity of BT200
- · Clinically evident bleeding



#### 1.3.2 Secondary Endpoints

#### Pharmacokinetic Endpoints:

- Measured concentration of BT200
- Derived PK parameters

#### 1.3.3 Exploratory Endpoints

- Immunogenicity Endpoint:
  - o ADAs against BT200
- Pharmacodynamic Endpoints:
  - o Platelet Function Analyzer (PFA-100®)
  - VWF:ristocetin co-factor assay (VWF:RiCo)
  - Multiplate electrode platelet aggregometer (ristocetin)
  - Enzyme-linked immunosorbent assay (ELISA) for unbound VWF-A1 domain (REAADS®)
- Biomarker Endpoints:
  - o VWF antigen and propeptide
  - Factor VIIIc activity (elagic acid activator)
  - o Activated partial thromboplastin time (aPTT) FS (elagic acid activator)
  - o Calibrated Automated Thrombogram (CAT) assay (Thrombinoscope®)

#### 1.4 Sample Size Calculation

As this study is exploratory and descriptive in nature, no inferential statistical testing was planned and therefore an exact sample size requirement cannot be specified. The number of NHVs planned to be included is expected to be sufficient to fulfill the study's objectives, but not excessive.

Part A: 80 NHVs; Part B: 16 NHVs; Part C: 8 NHVs; Part D: 8 NHVs (including NHVs who may have previously participated in Part A).

#### 1.5 Flowchart and Schedules of Assessments

Flowcharts for all study parts are provided in the Clinical Study Protocol (CSP), Section 'Study Diagram'.

ASSIGN DMB

#### Table 1: Study Procedures Part A (Weeks 1-14) (SAD)

| Visit | Screening | | | | | V1 | | | | V2 | V3 | V4 | V5 | V6 | V7 | | PK and<br>Immuno |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Tre | atment | | | | | | Post-tr | eatmen | t | | V8 | Sampling<br>Visits |
| Day | | | | | D0 | | | | D1 | D2 | D3 | D4 | D7 | D14 | D21 | D28 | D42, D56 |
| Time | | -1h | Oh | 0.5h | 1h | 4h | 8h | 14h | 24h | 48h | 72h | 96h | 168h | | | | |
| Time Window | D-28 to D-1 | ±59' | | ±15' | ±15' | ±30' | ±30' | ±120' | ±30' | ±2h | ±2h | ±2h | ±2h | ±1d | ±1d | ±1d | ±2d |
| Written Informed Consent | Х | | | | | | | | | | | | | | | | |
| Demographic Data | Х | | | | | | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | | | | | | |
| Admit to Inpatient Unit | | Х | | | | | | | | | | | | | | | |
| Inclusion / Exclusion Criteria | Х | Χ¹ | | | | | | | | | | | | | | | |
| Randomization | | Х | | | | | | | | | | | | | | | |
| Study Drug Administration | | | Х | | | | | | | | | | | | | | |
| Body Weight and Height <sup>2</sup> | Х | Х | | | | | | | | | | | | | | Х | |
| Physical Examination, Full | Х | | | | | | | | | | | | Х | | | Х | |
| Physical Examination, Brief | | Х | | | | | | | Х | Х | | | | Х | Х | | |
| Vital Signs (BP, HR, body temperature) | х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Cardiac Evaluation (12-lead ECG) | Х | Х | | | | | | | Х | | | | Х | | | Х | |
| Serology for HIV, hepatitis B, and hepatitis C | Х | | | | | | | | | | | | | | | | |
| Hematology | Х | Х | | | | Х | | | Х | Х | | | Х | Х | Х | Х | |
| Coagulation | Х | Х | | | | Х | | | Х | Х | | | Х | Х | Х | Х | |
| Clinical Chemistry | Х | Х | | | | Х | | | Х | Х | | | Х | Х | Х | Х | |
| Urinalysis <sup>3</sup> | Х | Х | | | | | | | Х | Х | | | Х | Х | Х | Х | |
| PK Assessments | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | <b>X</b> 4 |
| Immuno Assessments | | Х | | | | | | | | | | | | | | | <b>X</b> 4 |
| PD Assessments 5 | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |



| Visit | Screening | | | | | V1 | | | | V2 | V3 | V4 | V5 | V6 | V7 | | PK and |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Tre | atment | | | | | | Post-ti | reatment | t | | V8 | Immuno<br>Sampling<br>Visits |
| Day | | | | | D0 | | | | D1 | D2 | D3 | D4 | D7 | D14 | D21 | D28 | D42, D56 |
| Time | | -1h | Oh | 0.5h | 1h | 4h | 8h | 14h | 24h | 48h | 72h | 96h | 168h | | | | |
| Discharge from Inpatient<br>Unit | | | | | | | | | Х | | | | | | | | |
| Concomitant Medications /<br>Procedures | Х | | Ongoing | | | | | | | | | | | | | | |
| Adverse Events | Х | | | | | | | | Oı | ngoing | | | | | | | |

Abbreviations: '=minute(s); ADA=anti-drug antibody; BP=blood pressure; D=day; ECG=electrocardiogram; h=hour(s); HIV=human immunodeficiency virus; HR=heart rate; Immuno=immunogenicity; PD=pharmacodynamic(s); PK=pharmacokinetic(s); SAD=single ascending dose; V=visit

- 1. At -1h (ie, before BT200 injection) on Day 0, site personnel will perform a brief recheck of inclusion/exclusion criteria (excluding reassessments of laboratory parameters) to ensure that the subject remains eligible to participate in the study.
- 2. Body height will only be measured at Screening.
- 3. Dipstick urinalysis will be performed.
- 4. Late PK samples will be obtained at 6 and 8 weeks after the dose of study drug, whereas late immunogenicity samples will be obtained only at 8 weeks after the dose of study drug
- 5. PD assessments also include biomarker assays and an exploratory coagulation assay.

Note: Additional details regarding Part A laboratory blood sampling (hematology, coagulation, clinical chemistry, PK assessments, immunogenicity assessments, and PD assessments [including biomarker assays and an exploratory coagulation assay]) are provided in CSP Appendix 1: Laboratory Blood Sampling Supplement to Schedule of Assessments (Part A) and the laboratory manual.



Table 2: Study Procedures Part B Week 1 (MAD)

| Visit | Screening | | | | V | ′1 | | | | V2 | V3 | V4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | | | | | | | Treatmer | nt | | | | |
| | | | | | D0 | | | | D1 | D2 | D3 | D4 |
| Time | | -1h | Oh | 0.5h | 1h | 4h | 8h | 14h | 24h | 48h | 72h | 96h |
| Time Window | D-28 to D-1 | ±59' | | ±15' | ±15' | ±30' | ±30' | ±120' | ±30' | ±2h | ±2h | ±2h |
| Written Informed Consent | Х | | | | | | | | | | | |
| Demographic Data | Х | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | |
| Admit to Inpatient Unit | | Х | | | | | | | | | | |
| Inclusion / Exclusion Criteria | Х | Х | | | | | | | | | | |
| Randomization | | Х | | | | | | | | | | |
| Study Drug Administration <sup>1</sup> | | | Х | | | | | | | | | |
| Body Weight and Height <sup>2</sup> | Х | Х | | | | | | | | | | |
| Physical Examination, Full | Х | | | | | | | | | | | |
| Physical Examination, Brief | | Х | | | | | | | Х | | | Х |
| Vital Signs (BP, HR, body temperature) | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Cardiac Evaluation (12-lead ECG) | Х | Х | | | | | | | Х | | | |
| Serology for HIV, hepatitis B, and hepatitis C | Х | | | | | | | | | | | |
| Nasal swab screen for coronavirus | Х | | | | | | | | | | | |
| Hematology | Х | Х | | | | Х | | | Х | | | Х |
| Coagulation | Х | Х | | | | | | | Х | | | Х |
| Clinical Chemistry | Х | Х | | | | | | | Х | | | |
| Urinalysis <sup>3</sup> | Х | Х | | | | | | | Х | | | |
| PK Assessments | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Immunogenicity Assessments | | Х | | | | | | | | | | |
| PD Assessments <sup>4</sup> | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Discharge from Inpatient Unit 5 | | | | | | | | | Х | | | |



| Visit | Screening | | | | V | 1 | | | | V2 | V3 | V4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Day | | Treatment D1 D2 D3 D4 | | | | | | | | | | |
| | | | | | D0 | | | | D1 | D2 | D3 | D4 |
| Time | | -1h | Oh | 0.5h | 1h | 4h | 8h | 14h | 24h | 48h | 72h | 96h |
| Concomitant Medications / Procedures | Х | | | | | | Ongoing | | | | | • |
| Adverse Events | Х | | | | | | Ongoing | , | | | | |

Abbreviations: '=minute(s); ADA=anti-drug antibodies; BP=blood pressure; D=day; ECG=electrocardiogram; h=hour(s); HIV=human immunodeficiency virus; HR=heart rate; MAD=multiple ascending dose; PD=pharmacodynamic(s); PK=pharmacokinetic(s); V=visit

- 1. Study drug will be administered after all other study procedures for this visit have been completed.
- 2. Body height will only be measured at Screening.
- 3. Dipstick urinalysis will be performed.
- 4. PD assessments also include biomarker assays and an exploratory coagulation assay.
- 5. Based on the results from Part A, it may become apparent that the overnight stay and Hour 14 blood sample time point in Part B are superfluous. In this case, at the discretion of the Principal Investigator, the Hour 14 time point procedures may be omitted and the subjects discharged after the Hour 8 time point procedures have been completed.

Note: Additional details regarding Part B laboratory blood sampling (hematology, coagulation, clinical chemistry, PK assessments, immunogenicity assessments, and PD assessments [including biomarker assays and an exploratory coagulation assay]) are provided in CSP Appendix 2: Laboratory Blood Sampling Supplement to Schedule of Assessments (Part B) and the laboratory manual.



Table 3: Study Procedures Part B Weeks 2-12 (MAD)

| Visit | | V5-8 | | V9-11 | | PK and Immuno |
|---|---|---|---|---|---|---|
| | | Treatment | | Post-treatment | V12 | Sampling Visits |
| Day | | D 7, D14, D21, D28 | | D35, D42, D49 | D56 | D70, D84 |
| Time | -1h | 0h | 1h | 0h | 0h | ±2d |
| Time Window | ±59' | | ±30' | | | |
| Study Drug Administration | | Х | | | | |
| Body weight | Х | | | | х | |
| Physical Examination, Full | | | <b>X</b> <sup>1</sup> | | <b>X</b> <sup>1</sup> | |
| Physical Examination, Brief | Х | | х | Х | | |
| Vital Signs (BP, HR, body temperature) | Х | | х | Х | х | |
| Cardiac Evaluation (12-lead ECG) | Х | | | | х | |
| Hematology | Х | | | Х | х | |
| Coagulation | Х | | | Х | х | |
| Clinical Chemistry | Х | | | Х | х | |
| Urinalysis <sup>2</sup> | Х | | | Х | х | |
| PK Assessments | Х | | | Х | х | <b>X</b> <sup>3</sup> |
| Immuno Assessments | Х | | | | | <b>X</b> 3 |
| PD Assessments <sup>4</sup> | Х | | | Х | х | |
| Concomitant Medications / Procedures | Ongoing | | | | | |
| Adverse Events | Ongoing | | | | | |

Abbreviations: '=minute; BP=blood pressure; D=day; ECG=electrocardiogram; h=hour; HR=heart rate; Immuno=immunogenicity; MAD=multiple ascending dose; PD=pharmacodynamic(s); PK=pharmacokinetic(s); V=visit

- 1. Full physical examination only on Days 28 and 56.
- 2. Dipstick urinalysis will be performed.
- 3. Late PK samples will be obtained at 6 and 8 weeks after the last dose of study drug, whereas late immunogenicity samples will be obtained only at 8 weeks after the dose of study drug.
- 4. PD assessments also include biomarker assays and an exploratory coagulation assay.

Note: Additional details regarding Part B laboratory blood sampling (hematology, coagulation, clinical chemistry, PK assessments, immunogenicity assessments, and PD assessments [including biomarker assays and an exploratory coagulation assay]) are provided in CSP Appendix 2: Laboratory Blood Sampling Supplement to Schedule of Assessments (Part B) and the laboratory manual.



Table 4: Study Procedures Part C Weeks 1-9 (Desmopressin Challenge)

| Visit | Scr | V1 | | | | | | V2 | | | | | V3 | V4 | V5 | V6 | V7 | V8 | | PK and |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | _ | Treatm | ent | | | | | | | Post-tr | eatment | t | | V9 | Immuno<br>SaV |
| Day | | D -4 | | | | | D0 | | | | | D1 | D2 | D3 | D4 | D7 | D14 | D21 | D28 | D42, D56 |
| Time | | -96h | -1h | 0h | 0.5h | 1h | 2h | 3h | 4h | 8h | 14h | 24h | 48h | 72h | 96h | 168h | | | | |
| Time Window | D-28<br>to<br>D-5 | ±1h | ±59' | | ±15' | ±15' | ±15' | ±15' | ±30' | ±30' | ±120' | ±30' | ±2h | ±2h | ±2h | ±2h | ±1d | ±1d | ±1d | ±2d |
| Written Informed Consent | Х | | | | | | | | | | | | | | | | | | | |
| Demographic Data | Х | | | | | | | | | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | | | | | | | | | |
| Admit to Inpatient Unit | | | Х | | | | | | | | | | | | | | | | | |
| Inclusion / Exclusion<br>Criteria | Х | | X | | | | | | | | | | | | | | | | | |
| Randomization | | Х | | | | | | | | | | | | | | | | | | |
| Study Drug<br>Administration | | Х | | | | | | | | | | | | | | | | | | |
| Desmopressin<br>Administration | | | | Х | | | | | | | | | | | | | | | | |
| Body Weight and<br>Height <sup>1</sup> | Х | | Х | | | | | | | | | | | | | | | | х | |
| Physical Examination, Full | Х | | | | | | | | | | | | | | | Х | | | Х | |
| Physical Examination,<br>Brief | | | Х | | | | | | | | | Х | | | | | Х | Х | | |
| Vital Signs (BP, HR, body temperature) | Х | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | |
| Cardiac Evaluation<br>(12-lead ECG) | Х | | Х | | | | | | | | | Х | | | | Х | | | Х | |
| Serology for HIV,<br>hepatitis B, and<br>hepatitis C | Х | | | | | | | | | | | | | | | | | | | |
| Nasal swab screen for coronavirus | Х | | | | | | | | | | | | | | | | | | | |



| Visit | Scr | V1 | | | | | | V2 | | | | | V3 | V4 | V5 | V6 | V7 | V8 | | PK and |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | Treatm | ent | | | | | | | Post-tr | eatment | | | V9 | Immuno<br>SaV |
| Day | | D -4 | | | | | D0 | | | | | D1 | D2 | D3 | D4 | D7 | D14 | D21 | D28 | D42, D56 |
| Time | | -96h | -1h | 0h | 0.5h | 1h | 2h | 3h | 4h | 8h | 14h | 24h | 48h | 72h | 96h | 168h | | | | |
| Hematology | Х | Х | Х | | | X | Х | Х | Х | Х | | Х | | | | Х | | | Х | |
| Coagulation | Х | Х | Х | | | Х | Х | Х | Х | Х | | Х | | | | Х | | | Х | |
| Clinical Chemistry | Х | Х | Х | | | | | | | | | | | | | Х | | | | |
| Urinalysis <sup>2</sup> | Х | | Х | | | | | | | | | | | | | Х | | | Х | |
| PK Assessments | | Х | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | <b>X</b> 3 |
| Immuno Assessments | | Х | | | | | | | | | | | | | | | | | | <b>X</b> 3 |
| PD Assessments <sup>4</sup> | | Х | Х | | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Discharge from<br>Inpatient Unit | | | | | | | | | | | | Х | | | | | | | | |
| Concomitant<br>Medications /<br>Procedures | Х | | • | Ongoing | | | | | | | | | | | | | | | | |
| Adverse Events | Х | | | Ongoing | | | | | | | | | | | | | | | | |

Abbreviations: '=minute(s); BP=blood pressure; D=day; ECG=electrocardiogram; h=hour(s); HIV=human immunodeficiency virus; HR=heart rate; Immuno=immunogenicity; PD=pharmacodynamic(s); PK=pharmacokinetic(s); SaV=Sampling Visits; Scr=Screening; V=visit

- 1. Body height will only be measured at Screening.
- 2. Dipstick urinalysis will be performed.
- 3. Late PK samples will be obtained at 6 and 8 weeks after the dose of study drug, whereas late immunogenicity samples will be obtained only at 8 weeks after the dose of study drug.
- 4. PD assessments also include biomarker assays.

Note: Additional details regarding Part C laboratory blood sampling (hematology, coagulation, clinical chemistry, PK assessments, immunogenicity assessments, and PD assessments [including biomarker assays]) are provided in CSP Appendix 3: Laboratory Blood Sampling Supplement to Schedule of Assessments (Part C) and the laboratory manual.



Page 16 of 38

Table 5: Study Procedures Part D Weeks 1-8 (Relative Bioavailability)

| Visit | Screening | | | | | V1 | | | | V2 | V3 | V4 | V5 | V6 | V7 | | PK and |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Т | reatmer | nt | | | | | Post- | treatmer | nt | | V8 | Immuno<br>Sampling<br>Visits |
| Day | | | | | D | 00 | | | D1 | D2 | D3 | D4 | D7 | D14 | D21 | D28 | D42,<br>D56 |
| Time | | -1h | 0h | 0.5h | 1h | 4h | 8h | 14h | 24h | 48h | 72h | 96h | 168h | | | | |
| Time Window | D-28 to<br>D-1 | ±59' | | ±15' | ±15' | ±30' | ±30' | ±120' | ±30' | ±2h | ±2h | ±2h | ±2h | ±1d | ±1d | ±1d | ±2d |
| Written Informed Consent | Х | | | | | | | | | | | | | | | | |
| Demographic Data | Х | | | | | | | | | | | | | | | | |
| Medical History | Х | | | | | | | | | | | | | | | | |
| Admit to Inpatient Unit | | Х | | | | | | | | | | | | | | | |
| Inclusion / Exclusion Criteria | Х | Х | | | | | | | | | | | | | | | |
| Randomization | | Х | | | | | | | | | | | | | | | |
| Study Drug Administration | | | X <sup>4</sup> | | | | | | | | | | | | | | |
| Body Weight and Height <sup>1</sup> | Х | Х | | | | | | | | | | | | | | Х | |
| Physical Examination, Full | Х | | | | | | | | | | | | Х | | | Х | |
| Physical Examination, Brief | | Х | | | | | | | Х | | | | | Х | Х | | |
| Vital Signs (BP, HR, body temperature) | Х | Х | | Х | Х | Х | X | X | Х | Х | х | Х | Х | Х | Х | Х | |
| Cardiac Evaluation (12-lead ECG) | Х | Х | | | | | | | Х | | | | Х | | | Х | |
| Serology for HIV, hepatitis B, and hepatitis C | Х | | | | | | | | | | | | | | | | |
| Hematology | Х | Х | | | | | | | Х | | | | Х | | | Х | |
| Coagulation | Х | Х | | | | | | | Х | | | | Х | | | Х | |
| Clinical Chemistry | Х | Х | | | | | | | Х | | | | Х | | | Х | |
| Urinalysis | Х | X | | | | | | | Х | | | | Х | | | Х | |
| PK Assessments | | X | | Х | Х | Х | X | X | Х | Х | Х | Х | Х | Х | Х | Х | <b>X</b> <sup>2</sup> |
| Immuno Assessments | | Х | | | | | | | | | | | | | | | <b>X</b> <sup>2</sup> |
| PD Assessments <sup>3</sup> | | Х | | Х | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | |
| Discharge from Inpatient Unit | | | | | | | | | Х | | | | | | | | |

Adapted from:

STAT03\_A Statistical Analysis Plan Version 6.0, Effective Date 16-Feb-2018

Confidential and intellectual property of Assign DMB. No part of this document or its contents may be duplicated, referenced, published or otherwise disclosed in any form or by any means without prior written consent of Assign DMB.



| Visit | Screening | | | | | V1 | | | | V2 | V3 | V4 | V5 | V6 | V7 | | PK and |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Т | reatme | nt | | | | | Post- | treatmer | nt | | V8 | Immuno<br>Sampling<br>Visits |
| Day | | | | | D | 0 | | | D1 | D2 | D3 | D4 | D7 | D14 | D21 | D28 | D42,<br>D56 |
| Time | | -1h | 0h | 0.5h | 1h | 4h | 8h | 14h | 24h | 48h | 72h | 96h | 168h | | | | |
| Concomitant Medications / Procedures | Х | | | | | | | | ( | Ongoin | g | | | | | | |
| Adverse Events | Х | | | | | | | | ( | Ongoin | g | | | | | | |

Abbreviations: '=minute(s); ADAs=anti-drug antibodies; BP=blood pressure; D=day; ECG=electrocardiogram; h=hour(s); HIV=human immunodeficiency virus; HR=heart rate; Immuno=immunogenicity; PD=pharmacodynamic(s); PK=pharmacokinetic(s); V=visit

- 1. Body height will only be measured at Screening.
- 2. Late PK samples will be obtained at 6 and 8 weeks after the dose of study drug, whereas late immunogenicity samples will be obtained only at 8 weeks after the dose of study drug.
- 3. PD assessments also include biomarker assays.

Note: Additional details regarding Part D laboratory blood sampling (hematology, coagulation, clinical chemistry, PK assessments, immunogenicity assessments, and PD assessments [including biomarker assays]) are provided in Appendix 4: Laboratory Blood Sampling Supplement to Schedule of Assessments (Part D) and the laboratory manual.

4. Continuous IV infusion over 24 hours beginning at Time 0.



#### 2. GENERAL CONSIDERATIONS

#### 2.1 Rationale

BT200 is a PEGylated aptamer that binds to the A1 domain of human VWF and thereby inhibits VWF binding to platelet glycoprotein Ib (GP1b), the first step in the cascade of platelet-mediated thrombogenesis. Study BT200-01 is a Phase 1 FIH study designed to assess the human safety, tolerability, pharmacokinetics, and pharmacologic activity of BT200 in NHVs. In order to ensure the well-being of study subjects, some key safety measures have been incorporated into the design of this study, including use of sentinel pairs of subjects and an independent Data and Safety Monitoring Board (DSMB). In order to assess the effect of elevated VWF levels (as might be encountered in patients in the future) on the BT200 concentration-effect relationship,1 single-dose cohort of BT200 administered together with a secretagogue for VWF (desmopressin) will be included as Part C. Finally, in order to assess the relative bioavailability of BT200 via SC vs. IV administration, a single dose IV cohort will be included as Part D. Based upon the PK and PD data observed in Parts A, C, and D the nominal dose levels specified in Part B may be adjusted by means of a Substantial Amendment to this protocol prior to initiation of dosing therein.

#### 2.2 Conduct of Analysis

For Part A, B, C and D, a formal interim analysis is not planned. After all subjects have all visits of the respective study part performed, a topline analysis will be performed for Part A and D separately. Tables, Listings and Figures (TLFs) for the topline analysis can be found in Section 7.Topline analyses might be based on cleaned data for which no SDV was performed yet (due to Covid-19 pandemic, see Section 2.16). The final analysis of all study parts will be performed, when all study parts were fully SDVd, cleaned and once all external data are available and reconciled and the database is closed.

#### 2.3 Statistical Software and Quality Control

All statistical analyses will be performed using SAS® version 9.3 or higher. Tables, figures and data listings will be generated in Microsoft® Word® as well as PDF® format.

Quality control of SAS® programs will include a review of the whole process of result generation:

- Review of all analysis SAS® programs
- Review of SAS® log for errors, warnings and other notes that could indicate mistakes in the programs
- Review of all tables, listings and figures for completeness and correctness

#### 2.4 Applicable Standard Operating Procedures

The applicable Standard Operating Procedures (SOPs) of Assign DMB for this study are:

STAT03 Statistical Analysis Plan

STATO4 Interim Analysis

STAT05 Randomization and Unblinding

STAT06 Data Review Meeting



STATO7 Report Writing

SAS01 SAS General Principles

SAS04 Handling of Statistical Analyses

SASO6 CDISC\_ADaM

SASO7 CDSC\_Quality\_Control

#### 2.5 Blinding and Randomization

Subjects and study staff will be blinded to treatment assignment. Injections and infusions of BT200 or placebo will have a similar appearance. Unblinding for Part A and D will be performed after data entry for the respective study part is complete and database snapshot was performed for topline analysis. Unblinding for Part B and C will be performed after data entry for the respective study part is complete and database closure was performed.

In Part A, NHVs will be randomized to treatment with BT200 or placebo in a ratio of 3:1 in Cohorts 1 and 2, and in a ratio of 6:2 in Cohorts 3 to 10, except for the sentinel pair of subjects (1:1 ratio). For each of the remaining study parts (Parts B, C, and D), NHVs will be randomized to treatment with BT200 or placebo in a ratio of 6:2. If the site is able to recruit Asians in addition to Caucasians, a stratified randomization procedure will be performed according to Ethnicity. This stratification is not performed formally within the randomization list, but the sites instructed to not consider Asians for the sentinel pairs (to increase probability for Asians to not receive placebo).

#### 2.6 Descriptive Analyses

Descriptive analyses of continuous variables (summary statistics) will be described with the number of non-missing observations, arithmetic mean, standard deviation (±SD), median, quartiles (Q1 and Q3) and range (minimum and maximum).

Categorical variables (frequency statistics) will be described with the number of non-missing observations and percentages (%). Percentages will be calculated on the total number of non-missing observations, if not stated otherwise.

#### 2.7 Inferential Analyses

Two-sided 95% confidence intervals (Cls)will be calculated according to Altman will be calculated for certain safety tables (see Section 7).

#### 2.8 Center and Country Effect

Not applicable. This is a single-center study that will be conducted at the Department of Clinical Pharmacology, Medical University of Vienna at the Vienna General Hospital (AKH/MUW) in Vienna, Austria.

#### 2.9 Handling Missing Data

Generally, missing values will not be imputed and the analysis will be limited to observed values.



#### 2.10 Protocol Deviations

For Part A and D, a Blind Data Review Meeting (BDRM) will be conducted prior to database snapshot for topline analysis. For Part B and C the BDRM will be conducted prior the database closure. BDRMs will be conducted on all data to review protocol deviations, to discuss specific unforeseeable data issues, and to allocate the subjects to the analysis sets. During the BDRM, two classifications will be performed:

- 1. Protocol deviations will be classified as not relevant or relevant deviations, based on the potential influence on the PK and PD analysis. Relevant protocol violations will include the following but are not limited to:
  - Violations of major inclusion or exclusion criteria
  - Wrong treatment administration
  - Other protocol deviations with expected substantial influence on PK analysis
- 2. Protocol deviations will be classified as important or not important with respect to the GCP (E3) definition (i.e. important protocol deviations are a subset of protocol deviations that may significantly impact the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being).

Protocol deviation classifications will be made on a case by case decision in the BDRM. The associated decisions will be documented and approved in the BDRM Report.

Protocol violations classified as important and/or relevant will be described in the CSR (Clinical Study Report).

#### 2.11 Medical Coding

Adverse events, medical history and concomitant procedures will be coded using MedDRA. Concomitant medications will be coded using WHO Drug Dictionary. Details are defined in the Coding Guideline. The used dictionary versions will be indicated in the respective tables and listings.

#### 2.12 Analysis Populations

#### 2.12.1 Safety Population

The Safety Population will include all randomized NHVs who received at least 1 dose of BT200/placebo. Subjects will be analyzed according to the treatment that they actually received. The Safety Population will be used for all safety endpoints.

#### 2.12.2 Per-Protocol Population

The Per-Protocol (PP) Population will comprise all NHVs of the Safety Population, if the following criteria are additionally met:

- All of the major inclusion criteria, none of the major exclusion criteria are fulfilled.
- Absence of other relevant protocol violations such as wrong treatment received.

For each study part, a PP Population will be defined in the BDRM. The PP Population will represent the primary PK and PD analysis population.



#### 2.13 Subject Data Listings

All subjects in the database will be included in listings if not stated otherwise. Data listings will include the subject number as identifier (and parameter and/or visit if available) and will be sorted by Dose cohort, subject ID (and parameter and/or visit if available). Every listing contains the column treatment group.

#### 2.14 Columns in Tables

The following columns will be used for tables, if not stated otherwise:

- Part A: Pooled Placebo column (over all dose levels), Cohort 1 BT200, Cohort 2 BT200, Cohort 3 BT200, Cohort 4 BT200, Cohort 5 BT200, Cohort 6 BT200, Cohort 7 BT200, Cohort 8 BT200, Cohort 9 BT200 and Cohort 10 BT200.
- Part B:Pooled Placebo (over all dose levels), Cohort 13 BT200, Cohort 14 BT200 and Pooled BT200 (all subjects treated with BT200 over all dose levels).
- Part C: Cohort 12 BT200 and Placebo column.
- Part D: Cohort 11 BT200 and Placebo column.

In each analysis part, a column showing all subjects together will additionally used in the table summarizing the demographic information.

#### 2.15 Changes in the Conduct of the Study or Planned Analysis

No changes to the statistical analysis as compared to CSP are planned.

#### 2.16 Effect of Covid-19

Due to the Covid-19 pandemic no monitoring visits can be performed before database snapshot for topline analyses. Possible impact of Covid-19 pandemic and respective measures were discussed. Subject visits and time points will be partly affected by the pandemic. If visits can not be performed due to Covid-19 the visit will be documented as not performed in the eCFR with reason "COVID19". Drop-outs due to Covid-19 will be documented in the eCRF on the end of study page with reason "other" and specification "COVID19" as reason for early termination. No further effects are expected due to Covid-19. Statistical analysis will include a summary of drop-outs and early terminations due to Covid-19. In Part B and C, a screening for coronavirus by nasal swab testing will be performed at the screening visit. Subjects with positive coronavirus test will be excluded from the study. The results of the coronavirus screening will be tabulated and listed.

Unexpected Covid-19 effects (e.g. overviews on missing data, Covid-19 related protocol deviations, missed visits, visits out of time-window and changes in study processes) will be described in the Clinical Study Report.

#### OVERALL STUDY INFORMATION

Tables will be provided for the Safety Population, if not stated otherwise and selected tables will be repeated for the PP Population. The following information will be analyzed descriptively and corresponding details on the subject level will be provided in data listings:



- · Patient overview
- Screening failures
- Violated inclusion/exclusion criteria (will only be listed)
- Subjects by dose level and overall
- Study visit information (incl. Admission/Discharge Inpatient Unit information)
- Missed visits due to Covid-19 (will be listed only)
- End of study information (incl. drop-outs due to Covid-19)
- Protocol deviations
- Coronavirus screening (only applicable for Part B and C)

Specifications of Tables, Listings and Figures (TLFs) are provided in Section 7.

#### 4. BASELINE EVALUATION

Baseline data will be presented for Safety Population .

#### 4.1 Data Points

Data will be analyzed from the screening visit and the randomization visit (if applicable) The following information will be analyzed descriptively and corresponding details on the subject level will be provided in data listings:

- Demographics (including body height [cm] and body weight [kg], Body Mass Index (BMI) [kg/m²])
- Serology (will only be listed)
- Medical history overall and by SOC and PT
- Prior/Concomitant medications overall and by ATC level
- Prior/Concomitant procedures overall and by SOC and PT
- Childbearing-potential (will only be listed)

Vital signs, ECG and physical examination results will be analyzed in the safety section (see Section 6.4). Specifications of TLFs are provided in Section 7.

#### 4.2 Derivations and Definitions

- Medications stopped clearly prior to first study drug administration will be considered as prior medications, all other medications are considered to be concomitant. Medications with a missing or incomplete stop date where it cannot clearly be decided if the stop date was before or after Day 0 (Visit 1) will be considered as concomitant.
- Procedures stopped clearly prior to first study drug administration will be considered as prior procedures, all other procedures are considered to be concomitant. Procedures with a missing or incomplete stop date where it cannot clearly be decided if the stop date was before or after Day 0 (Visit 1) will be considered as concomitant.
- BMI [kg/m²] is defined as the weight [kg] divided by the square of the body height [m]



#### 5. PHARMACOKINETICS / PHARMACODYNAMICS / BIOMARKER / IMMUNOGENICITY

Pharmacodynamics, biomarker and immunogenicity analysis will be performed for the PP Population and the Safety Population.

#### 5.1 Pharmacokinetics

Pharmacokinetics analysis will be performed by CERTARA and are not described in this Statistical Analysis Plan.

#### 5.2 Pharmacodynamics

The following tables will be performed for PFA-100, VWF:RiCo [%], multiplate aggregometer and REAADS and corresponding details on the subject level will be provided in data listings:

- Absolute values by time point
- Absolute change from randomization by time point
- Relative change [%] from randomization by time point

The following figures will be provided for PFA-100, VWF:RiCo [%], multiplate aggregometer and REAADS separately:

- Absolute values by subject: For every subject separately, the time course over of the parameters mentioned above will be drawn, where the actual measurement time point since first dose will be shown on x-axis (hours) and the parameters values will be drawn on the y-axis.
- Absolute values by cohort: One graph will be drawn that includes the data of all cohorts. One line will be
  drawn per cohort, where the x-axis will show the planned time point of measurement (in hours) and the yaxis will show the mean value of the respective cohort incl. standard error. Measurements of all scheduled
  visits will be included, where the EOS visit will be treated as the last visit.

PD sampling results will be entered eCRF using a result specifier (i.e. <,  $\le$ , >,  $\ge$ ). For statistical analysis, values reported as <x, >x or  $\ge$ x will be analyzed as x. E.g. <300, <300 or  $\ge$ 300 will be analyzed as value 300.

Details are specified in Section 7.

#### 5.3 Biomarker

The following tables will be performed for VWF antigen [%], VWF propertide [mIU/mL], Factor VIIIc activity [%], aPTT FS [sec], Thrombin generation CAT assay (Thrombinoscope) [nM], Fibrin D-dimer [mIU/mL] and Prothrombin fragment F1.2 [mIU/mL]. Corresponding details on the subject level will be provided in data listings:

- Absolute values by time point
- Absolute change from randomization by time point
- Relative change [%] from randomization by time point

The following figures will be provided for VWF antigen [%], VWF propertide [mIU/mL], Factor VIIIc activity [%], aPTT FS [sec], Thrombin generation CAT assay (Thrombinoscope) [nM] and Fibrin D-dimer [mIU/mL] and Prothrombin fragment F1.2 [mIU/mL] separately:



- Absolute values by subject: For every subject separately, the time course over of the parameters mentioned above will be drawn, where the actual measurement time point will be shown on x-axis (hours) and the parameters values will be drawn on the y-axis.
- Absolute values by cohort: One graph will be drawn that includes the data of all cohorts. One line will be
  drawn per cohort, where the x-axis will show the planned time point of measurement (in hours) and the yaxis will show the mean value of the respective cohort incl. standard error. Measurements of all scheduled
  visits will be included, where the EOS visit will be treated as the last visit.

Details are specified in Section 7.

#### 5.4 Immunogenicity

The following tables will be produced for immunogenicity and corresponding details on the subject level will be provided in data listings:

ADA results (positive/negative/not reportable/NA) by time point

Details are specified in Section 7.

#### 6. SAFETY ANALYSIS

All analyses will be performed for the Safety Population. Data from unscheduled visits will only be listed. Data from scheduled visits and early termination visits will be tabulated.

#### 6.1 Extent of Exposure

Study drug administration will be listed.

For Part B, a cumulative dose level will be determined as the total amount of received study drug up to the current time point (loading dose and maintenance dose).

For Part C, Desmopressin administration will be listed additionally.

#### 6.2 Adverse Events and Bleeding Events

Adverse Events (AEs) are documented in the eCRF section "Adverse Events" and Bleeding Events in the eCRF section "Bleedings". AEs and bleeding events will be analyzed together.

#### 6.2.1 Data Points

The following tables will be generated:

AE and bleeding event overview (e.g. any AE or bleeding event, any severe AE or bleeding event, any related AE or bleeding event, any hemorrhage (MedDRA SMQ), all embolic and thrombotic events (SMQ), Embolic and thrombotic events, arterial (SMQ), Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous (SMQ), Embolic and thrombotic events, venous (SMQ))

- )
- AEs and bleeding events overall and by SOC and PT



- Related AEs and bleeding events overall and by SOC and PT
- Serious AEs and bleeding events overall and by SOC and PT
- Related serious AEs and bleeding events overall and by SOC and PT
- AEs and bleeding events by maximum severity
- Related AEs and bleeding events by maximum severity
- Serious AEs and bleeding events by maximum severity
- Related serious AEs and bleeding events by maximum severity
- AEs and bleeding events leading to permanently study drug discontinuation or leading to withdrawn from study
- Related AEs and bleeding events leading to permanently study drug discontinuation or leading to withdrawn from study
- Major bleeding events overall and by SOC and PT
- Total ISTH bleeding score (frequency table)
- Bleeding Assessment Score by symptom
- Maximum Bleeding Assessment Score
- AEs and bleeding events with missing assessments (will only be listed)

#### 6.2.2 Definitions and Derivations

- AEs and bleeding events are considered as "related" if the causality to study drug is reported as "related" or "possible".
- Tables showing AEs or bleeding events by causality, subjects will be counted only in the strongest relationship category but events will be counted in each category.
- In tables showing AEs or bleedings events by maximum severity, subjects will be counted only in the highest grading category but events will be counted in each category.
- An AE or bleeding event is considered as "leading to permanently study drug discontinuation" if "study drug
  permanently discontinued" is ticked for "action taken on study treatment".
- An AE or bleeding event is considered as "leading to withdrawal from study" if for "Other action taken", "withdrawn from study" is answered with "yes".
- Missing assessments contains missing seriousness, severity and/or causality
- The Total ISTH Bleeding Score will be calculated as the sum of bleeding assessment scores (documented
  in the eCRF) overall symptoms of a subject. If a subject experienced a symptom more than once, the event
  with the higher bleeding score will be used.
- The SMQ code for Hemorrhage is 20000038 Haemorrhages (SMQ) which consists of SMQ codes 20000039 "Haemorrhage terms (excl laboratory terms)" and 20000040 "Haemorrhage laboratory terms".
- The SMQ code for arterial embolic and thrombotic events is 20000082 "Embolic and thrombotic events, arterial (SMQ)".



- The SMQ code for vessel type unspecified and mixed arterial and venous embolic and thrombotic events is 20000083 "Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous (SMQ)".
- The SMQ code for venous embolic and thrombotic events is 20000084 "Embolic and thrombotic events, venous (SMQ)".

#### 6.3 Laboratory Parameters

Laboratory data from scheduled visits and early termination visits will be tabulated. Listings will additionally include results from unscheduled visits.

The following parameters will be assessed in the study and will be included in the statistical analysis:

- Hematology
  - o Hemoglobin
  - Hematocrit
  - Red blood cells
  - White blood cells
  - Lymphocytes
  - o Monocytes
  - Neutrophils
  - Eosinophils
  - Basophils
  - Platelets
  - Reticulocytes
- Coagulation
  - o Prothrombin time
- Clinical Chemistry
  - o Sodium
  - o Potassium
  - o Calcium
  - o Chloride
  - o Aspartate aminotransferase
  - Alanine aminotransferase
  - o Alkaline phosphatase
  - o Lactate dehydrogenase
  - o Gamma-glutamyltransferase
  - o Bilirubin
  - C-reactive protein
  - Blood Urea Nitrogen
  - Creatinine



- Glucose
- Urinalysis
  - Specific gravity
  - o pH
  - Leukocytes
  - Nitrite
  - Protein
  - o Glucose
  - Ketones
  - Urobilinogen
  - Bilirubin
  - Erythrocytes

Quantitative laboratory parameters (i.e., hematology, clinical chemistry, coagulation, pH, Specific Gravity) will be analyzed descriptively:

- Absolute values by parameter and time point (summary statistics)
- Absolute change from randomization by parameter and time point (summary statistics)
- Relative change from randomization by parameter and time point (summary statistics)
- Number of subjects with values above/below normal range by parameter and time point (frequency statistics)

Qualitative urinalysis parameters will be analyzed by tabulation of urinalysis result by parameter and time point (frequency statistics)

One set of data listings will show parameters outside normal range (hematology, coagulation, clinical chemistry, quantitative urinalysis parameters) and abnormal qualitative urinalysis values, respectively.

For every parameter, boxplots showing the absolute values by study day will be provided.

All parameters will be analyzed using the unit registered by study site in the eCRF. No unit conversion will be done.

#### 6.4 Other Safety Parameters

Other safety data from scheduled visits will be tabulated as described below. Listings will additionally include results from unscheduled visits or early termination visit.

Results from vital signs (systolic blood pressure [mmHg], diastolic blood pressure [mmHg], heart rate [beats/min], body temperature [C] and body weight [kg]) and ECG will be tabulated descriptively by:

- Absolute values by parameter and time points (summary statistics)
- Absolute changes from randomization by parameter and time points (summary statistics)
- Number of subjects with clinically relevant vital signs results by parameter and time point (frequency statistics)



- ECG Interpretation (normal/abnormal/abnormal, clinically relevant/abnormal, not clinically relevant) by time point (frequency statistics)
- Physical examination results (normal/abnormal) by body system and time point (frequency statistics)

Absolute values of vital signs parameters and continuous ECG parameters will be provided by time point. The x-axis will show the study day. A separate figure will be provided for every parameter.

Details are specified in Section 7.

### 7. LIST OF TABLES, DATA LISTINGS AND FIGURES

The x in the numbering of the TLFs below has to be replaced by 1 for Part A, 2 for Part B, 3 for Part C and 4 for Part D.



#### 7.1 List of Tables

| No | Topline<br>Analysis | Title | Content/Comment |
|---|---|---|---|
| Overall Study | | I<br>ion and Baseline Evaluation | |
| 14.x.1.1.1 | Yes | Patient Overview | <ul> <li>Number of subjects in Safety Population</li> <li>Number of subjects in PP Population</li> <li>Number of sentinel subjects (only applicable for Part A)</li> <li>Number of randomized subjects</li> <li>Screening of coronavirus (only applicable for Part B and C)</li> <li>Columns: Not randomized, column for each BT200 dose level and Placebo</li> </ul> |
| 14.x.1.1.2 | No | Number of Screening Failures and Reasons | One column for all subjects |
| 14.x.1.1.3 | No | Subjects by Visit (Safety Population) | -, |
| 14.x.1.1.4 | No | End of Study Information (Safety Population) | <ul> <li>Visit attendance status</li> <li>Primary reason for early termination</li> <li>Early terminations due to Covid-19</li> </ul> |
| 14.x.1.1.5 | No | Protocol Deviations (Safety Population) | <ul> <li>Any major protocol deviation</li> <li>Major protocol deviations by category</li> <li>Any minor protocol deviation</li> <li>Minor protocol deviations by category</li> </ul> |
| 14.x.1.1.6 | Yes | Demographic Information (Safety Population) | <ul> <li>Gender</li> <li>Age [years]</li> <li>Race</li> <li>Ethnicity</li> <li>Body height [cm]</li> <li>Body weight [kg]</li> <li>BMI [kg/m²] at screening</li> </ul> |
| 14.x.1.1.7 | No | Medical History Overall and by SOC and PT (Safety Population) | <ul><li>Any medical history</li><li>By SOC and PT</li></ul> |
| 14.x.1.1.8 | No | Prior Medications Overall and by ATC Level (Safety Population) | Any prior medication By ATC level |
| 14.x.1.1.9 | No | Concomitant Medications Overall and by ATC Level (Safety Population) | <ul><li>Any concomitant medication</li><li>By ATC level</li></ul> |
| 14.x.1.1.10 | No | Prior Procedures Overall and by SOC and PT (Safety Population) | <ul><li>Any prior procedures</li><li>By SOC and PT</li></ul> |
| 14.x.1.1.11 | No | Concomitant Procedures Overall and by SOC and PT (Safety Population) | <ul><li>Any concomitant procedures</li><li>By SOC and PT</li></ul> |



| 14.x.1.2.3- | No | Repeat tables 14.x.1.1.3-5 for PP Population |
|---|---|---|
| 14.x.1.2.5 | INO | Repeat tables 14.X.1.1.5-5 for FF Fopulation |
| | namics/R | I<br>Biomarker/Immunogenicity |
| 14.x.2.1.1 | Yes | Multiplate Aggregometer [U]: Absolute values by time |
| 14.7.2.1.1 | 165 | point (PP Population) |
| 14.x.2.1.2 | No | Multiplate Aggregometer [U]: Absolute change from |
| 14.7.2.1.2 | INO | randomization by time point (PP Population) |
| 14.x.2.1.3 | No | Multiplate Aggregometer [U]:Relative change [%] from |
| 17.7.2.1.3 | INO | randomization by time point (PP Population) |
| 14.x.2.1.4 | Yes | PFA-100 [sec]: Absolute values by time point (PP |
| 14.7.2.1.4 | 163 | Population) |
| 14.x.2.1.5 | No | PFA-100 [sec]: Absolute change from randomization |
| 14.7.2.1.0 | 110 | by time point (PP Population) |
| 14.x.2.1.6 | No | PFA-100 [sec]: Relative change [%] from |
| 11.7.12.11.0 | 110 | randomization by time point (PP Population) |
| 14.x.2.1.7 | Yes | REAADS: Absolute values by time point (PP |
| 11.7.2.1.7 | 100 | Population) |
| 14.x.2.1.8 | No | REAADS: Absolute change from randomization by |
| 11.7.2.1.0 | 110 | time point (PP Population) |
| 14.x.2.1.9 | No | REAADS: Relative change [%] from randomization by |
| 11/1/21/210 | 10 | time point (PP Population) |
| 14.x.2.1.10 | Yes | VWF:RiCo [%]: Absolute values by time point (PP |
| | | Population) |
| 14.x.2.1.11 | No | VWF:RiCo [%]: Absolute change from randomization |
| | | by time point (PP Population) |
| 14.x.2.1.12 | No | VWF:RiCo [%]: Relative change [%] from |
| | | randomization by time point (PP Population) |
| 14.x.2.1.13 | Yes | VWF antigen [%]: Absolute values by time point (PP |
| | | Population) |
| 14.x.2.1.14 | No | VWF antigen [%]: Absolute change from |
| | | randomization by time point (PP Population) |
| 14.x.2.1.15 | No | VWF antigen [%]: Relative change [%] from |
| | | randomization by time point (PP Population) |
| 14.x.2.1.16 | Yes | VWF propeptide [mIU/mL]: Absolute values by time |
| | | point (PP Population) |
| 14.x.2.1.17 | No | VWF propeptide [mIU/mL]: Absolute change from |
| | | randomization by time point (PP Population) |
| 14.x.2.1.18 | No | VWF propeptide [mIU/mL]: Relative change [%] from |
| | | randomization by time point (PP Population) |
| 14.x.2.1.19 | Yes | Factor VIIIc activity [%]: Absolute values by time point |
| | | (PP Population) |
| 14.x.2.1.20 | No | Factor VIIIc activity [%]: Absolute change from |
| 11 0101 | | randomization by time point (PP Population) |
| 14.x.2.1.21 | No | Factor VIIIc activity [%]: Relative change [%] from |
| 14 × 0 4 00 | Voc | randomization by time point (PP Population) |
| 14.x.2.1.22 | Yes | aPTT FS [sec]: Absolute values by time point (PP |
| 14 y 0 4 00 | No | Population) |
| 14.x.2.1.23 | INO | aPTT FS [sec]: Absolute change from randomization |
| 14 , 0 1 0 1 | No | by time point (PP Population) |
| 14.x.2.1.24 | No | aPTT FS [sec]: Relative change from randomization |
| 14.x.2.1.25 | Voc | by time point (PP Population) |
| 14.x.2.1.25 | Yes | Thrombin generation CAT assay [nM]: Absolute values by time point (PP Population) |
| | l | values by time point (FF Fobulation) |



| | | 1 |
|---|---|---|
| No | | |
| | change from randomization by time point (PP | |
| | Population) | |
| No | Thrombin generation CAT assay [nM]: Relative | |
| | change [%] from randomization by time point (PP | |
| Yes | | |
| No | | |
| INO | | |
| No | | |
| INO | | |
| Yes | | |
| No | | |
| No | Prothrombin fragment F1.2 [mIU/mL]: Relative | |
| | change [%] from randomization by time point (PP | |
| | Population) | |
| No | | |
| 110 | | |
| cic | 1 opalation | |
| | ate. | |
| | | T |
| Yes | AE and bleeding event overview (Safety Population) | <ul> <li>Any AE or bleeding event</li> <li>Any related AE or bleeding event</li> <li>Any severe AE or bleeding event</li> <li>Any related severe AE or bleeding event</li> <li>Any serious AE or bleeding event</li> <li>Any related serious AE or bleeding event</li> <li>Any Hemorrhage (MedDRA SMQ)</li> <li>Any AEs or bleeding events leading to permanently study drug discontinuation or leading to withdrawn from study</li> <li>Any related AEs or bleeding events leading to permanently study drug discontinuation or leading to withdrawn from study</li> <li>Any related AEs or bleeding events leading to permanently study drug discontinuation or leading to withdrawn from study</li> <li>(repeat contents for bleeding events)</li> <li>Any Hemorrhage Event</li> </ul> |
| | Yes No No No No No No Sis | change from randomization by time point (PP Population) No Thrombin generation CAT assay [nM]: Relative change [%] from randomization by time point (PP Population) Yes Fibrin D-dimer [mIU/mL]: Absolute values by time point (PP Population) No Fibrin D-dimer [mIU/mL]: Absolute change from randomization by time point (PP Population) No Fibrin D-dimer [mIU/mL]: Relative change [%] from randomization by time point (PP Population) Yes Prothrombin fragment F1.2 [mIU/mL]: Absolute values by time point (PP Population) No Prothrombin fragment F1.2 [mIU/mL]: Absolute change from randomization by time point (PP Population) No Prothrombin fragment F1.2 [mIU/mL]: Relative change [%] from randomization by time point (PP Population) No ADA results by time point (PP Population) No Repeat tables 14.x.2.1.1-14.x.2.1.34 for Safety Population |



| | | | <ul> <li>All embolic and thrombotic events (SMQ)</li> <li>Embolic and thrombotic events, arterial (SMQ)</li> <li>Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous (SMQ)</li> <li>Embolic and thrombotic events, venous (SMQ)</li> </ul> |
|---|---|---|---|
| 14.x.3.1.2 | Yes | AEs and bleeding events overall and by SOC and PT (Safety Population) | |
| 14.x.3.1.3 | Yes | Related AEs and bleeding events overall and by SOC and PT (Safety Population) | |
| 14.x.3.1.4 | Yes | Severe AEs and bleeding events overall and by SOC and PT (Safety Population) | |
| 14.x.3.1.5 | Yes | Related severe AEs and bleeding events overall and by SOC and PT (Safety Population) | |
| 14.x.3.1.6 | Yes | Serious AEs and bleeding events overall and by SOC and PT (Safety Population) | |
| 14.x.3.1.7 | Yes | Related serious AEs and bleeding events overall and by SOC and PT (Safety Population) | |
| 14.x.3.1.8 | Yes | AEs and bleeding events by maximum severity (Safety Population) | Incl. 2-sided 95% Cls |
| 14.x.3.1.9 | Yes | Related AEs and bleeding events by maximum severity (Safety Population) | Incl. 2-sided 95% Cls |
| 14.x.3.1.10 | Yes | Serious AEs and bleeding events by maximum severity (Safety Population) | Incl. 2-sided 95% Cls |
| 14.x.3.1.11 | Yes | Related serious AEs and bleeding events by maximum severity (Safety Population) | Incl. 2-sided 95% Cls |
| 14.x.3.1.12 | Yes | AEs and bleeding events leading to permanently study drug discontinuation or leading to withdrawn from study by SOC and PT (Safety Population) | |
| 14.x.3.1.13 | Yes | Related AEs and bleeding events leading to permanently study drug discontinuation or leading to withdrawn from study by SOC an PT (Safety Population) | |
| 14.x.3.1.14 | Yes | Bleeding Events by SOC and PT (Safety population) | Incl. 2-sided 95% CI |
| 14.x.3.1.15 | Yes | Major bleeding events overall and by SOC and PT (Safety Population) | |
| 14.x.3.1.16 | Yes | Total ISTH Bleeding Score (Safety Population) | |
| 14.x.3.1.17 | Yes | Bleeding Assessment Score by Symptom (Safety Population) | |
| 14.x.3.1.18 | Yes | Maximum Bleeding Assessment Score (Safety Population) | |
| Laboratory p | | | |
| 14.x.3.1.19 | Yes | Hematology and Coagulation: Absolute values by time point (Safety Population) | |
| 14.x.3.1.20 | Yes | Hematology and Coagulation: Absolute change from randomization by time point (Safety Population) | |
| 14.x.3.1.21 | Yes | Hematology and Coagulation: Relative change from randomization by time point (Safety Population) | |



| 14.x.3.1.22 | Yes | Hematology and Coagulation: Subjects outside | |
|---|---|---|---|
| | | normal range by time point (Safety Population) | |
| 14.x.3.1.23 | Yes | Clinical Chemistry: Absolute values by time point | |
| | | (Safety Population) | |
| 14.x.3.1.24 | Yes | Clinical Chemistry: Absolute change from | |
| | | randomization by time point (Safety Population) | |
| 14.x.3.1.25 | Yes | Clinical Chemistry: Relative change from | |
| 11 0100 | | randomization by time point (Safety Population) | |
| 14.x.3.1.26 | Yes | Clinical Chemistry: Subjects outside normal range by | |
| 4424.07 | \/ | time point (Safety Population) | |
| 14.x.3.1.27 | Yes | Quantitative Urinalysis: Absolute values by time point | |
| 14.x.3.1.28 | Yes | (Safety Population) Quantitative Urinalysis: Absolute change from | |
| 14.3.3.1.20 | 165 | randomization by time point (Safety Population) | |
| 14.x.3.1.29 | Yes | Quantitative Urinalysis: Relative change from | |
| 14.7.3.1.29 | 163 | randomization by time point (Safety Population) | |
| 14.x.3.1.30 | Yes | Quantitative Urinalysis: Subjects outside normal | |
| 1.7.3.1.30 | 1.00 | range by time point (Safety Population) | |
| 14.x.3.1.31 | Yes | Qualitative Urinalysis by time point (Safety | |
| | | Population) | |
| 14.x.3.1.32 | Yes | Vital Signs: Absolute values by time point (Safety | systolic blood pressure |
| | | Population) | [mmHg] |
| | | | diastolic blood pressure |
| | | | [mmHg] |
| | | | heart rate [beats/min] |
| | | | body temperature [C] |
| | | | body weight [kg] |
| 14.x.3.1.33 | Yes | Vital Signs: Absolute change from randomization by | 3 8 1 63 |
| | | time point (Safety Population) | |
| | | | Content see Table 14.x.3.1.32 |
| 14.x.3.1.34 | Yes | Subjects with clinically relevant vital signs by time | |
| | | point (Safety Population) | Content see Table 14.x.3.1.32 |
| 14.x.3.1.35 | Yes | ECG: Absolute values by time point (Safety | • PQ [ms] |
| | | Population) | QRS [ms] |
| | | | • QT [ms] |
| | | | QTcF [ms] |
| | | | <ul> <li>P [ms]</li> </ul> |
| | | | • RR [ms] |
| | | | • PP [ms] |
| | | | P [degree] |
| | | | QRS [degree] |
| | | | T [degree] |
| 14.x.3.1.36 | Yes | ECG: Absolute change from randomization by time | |
| | | point (Safety Population) | Content see Table 14.x.3.1.35 |
| 4424.27 | | Subjects with clinically relevant ECG values by time | |
| 14.x.3.1.37 | Yes | | |
| | | point (Safety Population) | Content see Table 14.x.3.1.35 |
| 14.x.3.1.37 | | | Content see Table 14.x.3.1.35 • normal |
| | | point (Safety Population) | |
| | | point (Safety Population) | normal |
| | | point (Safety Population) | <ul><li>normal</li><li>abnormal</li><li>abnormal, clinically relevant</li></ul> |
| | | point (Safety Population) | <ul> <li>normal</li> <li>abnormal</li> <li>abnormal, clinically relevant</li> <li>abnormal, not clinically</li> </ul> |
| 14.x.3.1.38 | Yes | point (Safety Population) ECG Interpretation by time point (Safety Population) | <ul><li>normal</li><li>abnormal</li><li>abnormal, clinically relevant</li></ul> |
| | | point (Safety Population) ECG Interpretation by time point (Safety Population) Physical Examination results by body system and | <ul> <li>normal</li> <li>abnormal</li> <li>abnormal, clinically relevant</li> <li>abnormal, not clinically</li> </ul> |
| 14.x.3.1.38 | Yes | point (Safety Population) ECG Interpretation by time point (Safety Population) | <ul> <li>normal</li> <li>abnormal</li> <li>abnormal, clinically relevant</li> <li>abnormal, not clinically relevant</li> </ul> |



# 7.2 List of Data Listings

| No | Topline<br>Analysis | Title | Content/Comment |
|---|---|---|---|
| Overall Study | | n and Baseline Evaluation | |
| 16.2.x.1.1 | No | Analysis Population Details | Actual dose cohort, Randomized dose cohort, Subject number, Sentinel (only applicable for Part A), Randomization performed, Date of randomization, Time of randomization, Reason not randomized, Safety Population, Reason not in Safety Population, PP Population, Reason not in PP Population |
| 16.2.x.1.2 | No | Screening Failures with Reasons | Subject number, Informed consent date,<br>Subject's withdrawal of consent, In/Ex<br>criterion fulfilled, Adverse event, Other,<br>Specification other reason |
| 16.2.x.1.3 | No | Violated Entry Criteria | Subject number, Visit, Criterion ID not met, Criterion description |
| 16.2.x.1.4 | No | Visit Information and Admission/Discharge<br>Inpatient Unit | Dose cohort, Subject number, Visit, Reason for unscheduled visit, Visit/Admission/Discharge date, Visit/Admission/Discharge time, Reason visit not performed, Reason outside time window, Specification other reason, Age |
| 16.2.x.1.5 | No | Missed Visits due to Covid-19 | Dose cohort, Subject number, Visit,<br>Reason for unscheduled visit, Visit date,<br>Visit time, Reason visit not performed,<br>Reason outside time window, Age |
| 16.2.x.1.6 | No | Protocol Deviations | Dose cohort, Subject number, PD category, Classification, Reason for classification, PD description |
| 16.2.x.1.7 | Yes | Study End Information | Dose cohort, Subject number, Visit attendance status, Date of discontinuation, Primary reason for early termination, Specification other reason, Reason for recommended withdrawal, Death date, Primary cause of death |
| 16.2.x.1.8 | Yes | Drop-outs due to Covid-19 | Dose cohort, Subject number, Visit attendance status, Date of discontinuation, Primary reason for early termination, Specification other reason, Reason for recommended withdrawal, Death date, Primary cause of death |
| 16.2.x.1.9 | Yes | Demographic Data | Dose cohort, Subject number, Subject rescreened (only applicable for Part D), Subject number in Part A (only applicable for Part D), Date of informed consent, Year of birth, Age [years], Gender, Childbearing potential, Reason no childbearing potential, Specification other reason childbearing potential, Race, Specification other race, Ethnicity, Blood type, Rhesus factor, Body weight [kg] at |



| Screening for coronavirus by nasal swab Dose cohort, Subject number, Confection, Priser and Servicens of the study end Screening for coronavirus by nasal swab Dose cohort, Subject number, Confection, Priser and Servicens of the study end Screening for coronavirus by nasal swab Dose cohort, Subject number, Nedication, Therapy, ATC Level 2, ATC Level 3, Start date, End date, Ongoing at study end, Dose, Dose Unit, Dose Form, Frequency, Route, Indication category, prior/concomitant Dose cohort, Subject number, Procedure, Scr. Pr. Start date, End date, Ongoing at study end, Indication category, Indication, prior/concomitant Dose cohort, Subject number, Procedure, Scr. Pr. Start date, End date, Ongoing at study end, Indication category, Indication, prior/concomitant Dose cohort, Subject number, Visit, Serology sample collected, Reason not collected. Collection date, Collection time, Test name, Result, Not done Dose cohort, Subject number, Scr. Pharmacodynamics/Blomarker/Immunogenicity Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not collected, Collection time, Result Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result Specification, Result, Unit, Absolute Change, Relative Change % Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result Specification, Result, Unit, Absolute Change, Relative Change % Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change % Dose cohort, Subject number, Visit, Parameter, Sesult, Unit, Absolute Change, Relative Change, Rela | | _ | | |
|---|---|---|---|---|
| 16.2.x.1.10 No Medical History Dose cohort, Subject number, Condition, SC, PT, Start date, End date, Ongoing at study end Dose cohort, Subject number, Condition, SC, PT, Start date, End date, Ongoing at study end Dose cohort, Subject number, Medication/Therapy, ATC Level 2, ATC Level 3, Start date, End date, Ongoing at study end, Dose, Dose Dose Intil, Dose Form, Frequency, Route, Indication category, prior/concomittant | | | | screening, Body Height [cm], BMI [kg/m²] |
| SOC. PT. Start date, End date, Ongoing at study end | | | | |
| Study end Dose cohort, Subject number, Medication/Therapy, ATC Level 2, ATC Level 3, Start date, End date, Onglong at Study end, Dose, Dose Unit, Dose Form, Frequency, Route, Indication category, prior/concomitant | 16.2.x.1.10 | No | Medical History | Dose cohort, Subject number, Condition, |
| 16.2.x.1.11 No Concomitant Medications Dose cohort, Subject number, Medication/Therapy, ATC Level 2, ATC Level 3, Start date, End date, Ongoing at study end, Dose, Dose Unit, Dose Form, Frequency, Route, Indication category, prior/concomitant of Dose cohort, Subject number, Procedure, SOC, PT, Start date, End date, Ongoing at study end, Indication category, Indication, prior/concomitant Dose cohort, Subject number, Procedure, SOC, PT, Start date, End date, Ongoing at study end, Indication category, Indication, prior/concomitant Dose cohort, Subject number, Visit, Serology sample collected, Reason not collected, Collection date, Collecti | | | | SOC, PT, Start date, End date, Ongoing at |
| Medication/Therapy, ATC Level 2, ATC Level 3, Start date, End date, Ongoing at study end, Dose, Dose Unit, Dose Form, Frequency, Route, Indication category, prior/concomitant 16.2.x.1.12 | | | | study end |
| Medication/Therapy, ATC Level 2, ATC Level 3, Start date, End date, Ongoing at study end, Dose, Dose Unit, Dose Form, Frequency, Route, Indication category, prior/concomitant 16.2.x.1.12 | 16.2.x.1.11 | No | Concomitant Medications | Dose cohort, Subject number, |
| Level 3, Start date, End date, Ongoing at study end, Dose, Dose Unit, Dose Form, Frequency, Route, Indication category, prior/concomitant 16.2.x.1.12 No Concomitant Procedures Dose cohort, Subject number, Procedure, SOC, PT, Start date, End date, Ongoing at study end, Indication category, Indication, prior/concomitant 16.2.x.1.13 No Serology Dose cohort, Subject number, Visit, Serology sample collected, Reason not collected, Collection date, Collection time, Test name, Result, Not done 16.2.x.1.14 No Screening for coronavirus by nasal swab testing (only applicable for Part B and C) Pharmacodynamics/Biomarker/Immunogenicity 16.2.x.2.1 Yes Pharmacodynamics Results Dose cohort, Subject number, Sample collected, Collection date, Collection time, Result number, Sample taken, Reason not once of the collected of the collection time, Ave, Stdey, Cv%, Reported Result 16.2.x.2.2 Yes Additional Biomarker Results Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change (%) 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change (%) 16.2.x.3.1.1 Yes Study Drug Administration Dose level, Study drug administration End Time, Administration End Time, Location, Obse level, Study drug administered as, Reason not administered, Administration performed accor | | | | |
| Study end, Dose, Dose Unit, Dose Form, Frequency, Route, Indication category, prior/concomitant | | | | |
| Frequency, Route, Indication category, prior/concomitant | | | | |
| Prior/Concomitant | | | | |
| 16.2.x.1.12 No Concomitant Procedures Dose cohort, Subject number, Procedure, SOC, PT, Start date, End date, Ongoing at study end, Indication category, Indication, prior/concomitant | | | | |
| SOC, PT, Start date, End date, Ongoing at study end, indication category, indication, prior/concomitant indication category, indication, prior/concomitant of the prior concomitant in the prior collected, Collection date, Collection time, Test name, Result, Not done in the prior control subject number, Sample collected, Reason not collected, Collection date, Collection time, Result in the prior collected, Collection date, | 16 2 v 1 12 | No | Concomitant Procedures | |
| Study end, Indication category, Indication, prior/concomitant | 10.2.3.1.12 | INO | Concomitant Frocedures | The state of the s |
| Prior/concomitant Dose cohort, Subject number, Visit, Serology sample collected, Reason not collected, Collection date, Collection time, Test name, Result, Not done | | | | |
| 16.2.x.1.13 | | | | |
| Serology sample collected, Reason not collected, Collection date, Collection, Cher Location, Dose level, Study drug administration Start Date, Administration End Time, Administration End Time, Location, Other Location, Dose level, Study drug administration Start Date, Administration End Time, Administration End Time, Administration End Time, Inc. Date, Administration Start Date, Administration Start Date, Administration End Time, End Date, Administration End Time, End Date, Administration End Time, End Date, E | | | | |
| Collected, Collection date, Collection time, Test name, Result, Not done | 16.2.x.1.13 | No | Serology | The state of the s |
| time, Test name, Result, Not done | | | | Serology sample collected, Reason not |
| 16.2.x.2.14 No Screening for coronavirus by nasal swab testing (only applicable for Part B and C) Collection date, Collection time, Result | | | | collected, Collection date, Collection |
| testing (only applicable for Part B and C) Collected, Reason not collected, Collection time, Result Pharmacodynamics/Biomarker/Immunogenicity 16.2.x.2.1 Yes Pharmacodynamics Results Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.2 Yes Biomarker Results Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.2 Yes Additional Biomarker Results Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Nominal Day, Collection date, Collection time, Ave, Stdey, Cv%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administration Start Date, Administration Start Time, Administration Performed according to protocol, Cumulative dose level (only applicable for Part B) Dose cohort, Subject number, Desmopressin administration Start Date, Administration Start Time, Administration Start Time, Administration Start Time, Administration End Time, Administration End Time, Desmopressin administration End Time, Administration End Time, Desmopressin Administration End Time, Administration End Time, Desmopressin Administration End Time, De | | | | time, Test name, Result, Not done |
| testing (only applicable for Part B and C) Collected, Reason not collected, Collection time, Result Pharmacodynamics/Biomarker/Immunogenicity 16.2.x.2.1 Yes Pharmacodynamics Results Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.2 Yes Biomarker Results Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.2 Yes Additional Biomarker Results Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Nominal Day, Collection date, Collection time, Ave, Stdey, Cv%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administration Start Date, Administration Start Time, Administration Performed according to protocol, Cumulative dose level (only applicable for Part B) Dose cohort, Subject number, Desmopressin administration Start Date, Administration Start Time, Administration Start Time, Administration Start Time, Administration End Time, Administration End Time, Desmopressin administration End Time, Administration End Time, Desmopressin Administration End Time, Administration End Time, Desmopressin Administration End Time, De | 16.2.x.1.14 | No | Screening for coronavirus by nasal swab | |
| Collection date, Collection time, Result | | | | , , |
| Pharmacodynamics/Biomarker/Immunogenicity | | | terring (erri) approximate and a since of | |
| 16.2.x.2.1 Yes | Pharmacodyn | amics/Bio | <br>omarker/Immunogenicity | |
| Sampling Date/Time, Sample taken, Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change, Relative Change [%] 16.2.x.2.2 Yes Biomarker Results Dose cohort, Subject number, Visit, Sampling Date/Time, Sample taken, Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.2 Yes Additional Biomarker Results Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Nominal Day, Collection date, Collection time, Ave, Stdev, CV%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered, Study drug administered, Study drug administered, Study drug administered, Study drug administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Visit, Study drug administration End Time, Administration For Part B) Dose cohort, Subject number, Visit, Study drug administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Time, A | | | | Dose cohort Subject number Visit |
| Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] | 10.2.7.2.1 | 163 | Thatmacodynamics Results | |
| Specification, Result, Unit, Absolute Change, Relative Change [%] | | | | |
| Change, Relative Change [%] | | | | |
| 16.2.x.2.2 Yes | | | | |
| Sampling Date/Time, Sample taken, Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.2 Yes Additional Biomarker Results Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Nominal Day, Collection date, Collection time, Ave, Stdev, CV%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered, Study drug administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administered ose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Dose cohort, Subject number, Desmopressin administration Start Date, Administration Start Date, Administration Start Date, Administration Start Date, Administration Start Date, Administration Start Time, Administration End Time, Desmopressin administration Start Date, Administration Start Time, Administration End Time, Desmopressin administration Start Date, Administration End Time, Desmopressin administration Start Date, Administration End Time, Desmopressin administration Start Date, Administration End Time, Desmopressin administration Start Date, Administration End Time, Administration End Time, Desmopressin Admi | | | | |
| Reason not done, Test, Result specification, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.2 Yes Additional Biomarker Results Dose cohort, Subject number, Visit, Parameter, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Nominal Day, Collection date, Collection time, Ave, Stdev, CV%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered, Study drug administered, Study drug administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administered ose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration Start Date, Administration Start Time, Administration Start Date, Administration Start Time, Administration Start Date, Administration Start Time, Administration End Time, Incomplete Complete Compl | 16.2.x.2.2 | Yes | Biomarker Results | The state of the s |
| Specification, Result, Unit, Absolute Change, Relative Change [%] | | | | Sampling Date/Time, Sample taken, |
| Change, Relative Change [%] 16.2.x.2.2 Yes | | | | Reason not done, Test, Result |
| Additional Biomarker Results | | | | specification, Result, Unit, Absolute |
| Additional Biomarker Results | | | | Change, Relative Change [%] |
| Parameter, Result, Unit, Absolute Change, Relative Change [%] 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Nominal Day, Collection date, Collection time, Ave, Stdev, CV%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered, Study drug administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | 16.2.x.2.2 | Yes | Additional Biomarker Results | |
| Change, Relative Change [%] 16.2.x.2.3 No | | | | |
| 16.2.x.2.3 No ADA Results Dose cohort, Subject number, Nominal Day, Collection date, Collection time, Ave, Stdev, CV%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered as, Reason not administered, Administration Start Date, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Time, Administration End Date, Administration Start Time, Administration End Date, Administration End Time, | | | | |
| Day, Collection date, Collection time, Ave, Stdev, CV%, Reported Result Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered as, Reason not administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Time, | 16 2 v 2 3 | No | ADA Poculto | |
| Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered as, Reason not administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | 10.2.3.2.3 | INO | ADA Nesuits | , , |
| Safety Analysis 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered as, Reason not administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | |
| 16.2.x.3.1.1 Yes Study Drug Administration Dose cohort, Subject number, Visit, Study drug administered, Study drug administered as, Reason not administered, Administration Start Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | 0.6.4.4 | | | Staev, CV%, Reported Result |
| drug administered, Study drug administered as, Reason not administered as, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | |
| administered as, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | 16.2.x.3.1.1 | Yes | Study Drug Administration | |
| administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | |
| Administration Start Time, Administration End Date, Administration End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | , and the second |
| End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | administered, Administration Start Date, |
| End Date, Administration End Time, Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | Administration Start Time, Administration |
| Location, Other Location, Dose level, Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | |
| Study drug administration performed according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | |
| according to protocol, Cumulative dose level (only applicable for Part B) 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | | | | |
| Level (only applicable for Part B) 16.2.x.3.1.2 Yes | | | | |
| 16.2.x.3.1.2 Yes Desmopressin Administration (only applicable for Part C) Dose cohort, Subject number, Desmopressin administered, Reason not administered, Administration Start Date, Administration End Date, Administration End Time, | | | | |
| applicable for Part C) Desmopressin administered, Reason not administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | 16 2 v 2 1 2 | Vec | Desmonressin Administration (only | |
| administered, Administration Start Date, Administration Start Time, Administration End Date, Administration End Time, | 10.2.X.3.1.2 | res | | |
| Administration Start Time, Administration End Date, Administration End Time, | | | applicable for Part C) | · |
| End Date, Administration End Time, | | | | |
| | 1 | i | | Administration Start Time, Administration |
| Administration dose (ug) | | | | · |
| / Administration asso (48) | | | | End Date, Administration End Time, |
| | | | applicable for Part C) | administered, Administration Start Date, |
| | | | | · |



| 16.2.x.3.2 | Yes | Adverse Events (Part I) | Dose cohort, Subject number, Source, |
|---|---|---|---|
| | | | Term, SOC, PT, Start date, Start time, |
| | | | Serious, Serious Criteria, Severity, |
| | | | Causality to study treatment, Causality to |
| | | | desmopressin (only applicable for Part C) |
| 16.2.x.3.3 | Yes | Adverse Events (Part II) | Dose cohort, Subject number, AE Term, |
| 10121/11010 | | Thaveree Events (Fareil) | Action taken on study treatment, Action |
| | | | taken on desmopressin (only applicable |
| | | | for Part C), Other action taken, |
| | | | Specification other action taken, |
| | | | Outcome, Recovering date, recovering |
| | | | time, Ongoing at final examination |
| 16.2.x.3.4 | Yes | Serious Adverse Events (Part I) | See Listing 16.x.3.1 |
| 16.2.x.3.5 | | , , | _ |
| | Yes | Serious Adverse Events (Part II) | See Listing 16.x.3.2 |
| 16.2.x.3.6 | Yes | Haemorrhage terms (SMQ) (Part I) | See Listing 16.x.3.1 |
| 16.2.x.3.7 | Yes | Haemorrhage terms (SMQ) (Part II) | See Listing 16.x.3.2 |
| 16.2.x.3.8 | Yes | Embolic and thrombotic events, arterial (SMQ) (Part I) | See Listing 16.x.3.1 |
| 16.2.x.3.9 | Yes | Embolic and thrombotic events, arterial | See Listing 16.x.3.2 |
| | | (SMQ) (Part II) | |
| 16.2.x.3.10 | Yes | Embolic and thrombotic events, vessel type | See Listing 16.x.3.1 |
| | | unspecified and mixed arterial and venous | _ |
| | | (SMQ) (Part I) | |
| 16.2.x.3.11 | Yes | Embolic and thrombotic events, vessel type | See Listing 16.x.3.2 |
| | | unspecified and mixed arterial and venous | S |
| | | (SMQ) (Part II) | |
| 16.2.x.3.12 | Yes | Embolic and thrombotic events, venous | See Listing 16.x.3.1 |
| | | (SMQ) (Part I) | |
| 16.2.x.3.13 | Yes | Embolic and thrombotic events, venous | See Listing 16.x.3.2 |
| | | (SMQ) (Part II) | |
| 16.2.x.3.14 | No | Adverse Events with missing assessments | See Listing 16.x.3.1 |
| 100 015 | | (Part I) | |
| 16.2.x.3.15 | No | Adverse Events with missing assessments (Part II) | See Listing 16.x.3.2 |
| 16.2.x.3.16 | Yes | Additional Assessments for Bleeding Events | Dose cohort, Subject number, Bleeding |
| 10.2.3.10 | 165 | Additional Assessments for Dieeding Events | event, Bleeding event verbatim, Start |
| | | | date, Start time, Bleeding Assessment |
| | | | Score, ISTH clinical relevant major |
| | | | bleeding, Major bleeding criteria, ISTH |
| | | | clinical relevant non-major bleeding, Non- |
| | | | major bleeding criteria, End date, End |
| 100 017 | | | time |
| 16.2.x.3.17 | Yes | Hematology and Coagulation Values | Dose Level, Subject number, Parameter, |
| | | Outside Normal Range | Visit, Lab performed, Reason not |
| | | | performed, Collection date, Collection |
| | | | time, same as visit/admission/discharge |
| | | | date, Test, Result, Unit, not done, Reason |
| | | | not done, Outside laboratory limits, Lower |
| | | | limit, Upper limit, Clinically relevant |
| 16.2.x.3.18 | Yes | Clinical Chemistry Values Outside Normal<br>Range | See Listing 16.x.3.9 |
| | l | Quantitative Urinalysis Values Outside | See Listing 16.x.3.9 |
| 162 x 3 10 | LINO | r Sasariatativo Simialvala valuE3 VULSIUE | TOOU LIGHTING TO.A.U.U |
| 16.2.x.3.19 | No | Normal Range | |
| 16.2.x.3.19<br>16.2.x.3.20 | No | | Dose level, Subject number, Parameter, |
| | | Normal Range | |



| | | | time, same as visit/admission/discharge date, Result, not done, Reason not done, Clinically relevant |
|---|---|---|---|
| 16.2.x.3.21 | No | Vital Signs | Dose level, Subject number, Visit, Vital signs collection, Reason not collected, Collection date, Collection time, same as visit/admission/discharge date, Test, Result, Clinically relevant, not done |
| 16.2.x.3.22 | No | ECG | Dose level, Subject number, Visit, ECG performed, Reason not performed, Date, Time, Same as visit/admission/discharge date, Test, Result, Abnormal, Clinically relevant, not analyzed/not available |
| 16.2.x.3.23 | No | Physical Examination | Dose level, Subject number, Visit, Extent of physical examination, Examination performed, Reason not performed, Examination Date, Examination Time, same as visit/admission/discharge date, Body system, Result, Specification other body system |

# 7.3 List of Figures

| No | Topline | Title | Content/Comment |
|---|---|---|---|
| | Analysis | | |
| PD / Biomar | ker | | |
| 14.x.2.1.29 | Yes | Multiplate Aggregometer [U]: Absolute values by subject (PP Population) | |
| 14.x.2.1.30 | Yes | Multiplate Aggregometer [U]: Absolute values by cohort (PP Population) | |
| 14.x.2.1.31 | Yes | PFA-100 [sec]: Absolute values by subject (PP Population) | |
| 14.x.2.1.32 | Yes | PFA-100 [sec]: Absolute values by cohort (PP Population) | |
| 14.x.2.1.33 | Yes | REAADS: Absolute values by subject (PP Population) | |
| 14.x.2.1.34 | Yes | REAADS: Absolute values by cohort (PP Population) | |
| 14.x.2.1.35 | Yes | VWF:RiCo [%]: Absolute values by subject (PP Population) | |
| 14.x.2.1.36 | Yes | VWF:RiCo [%]: Absolute values by cohort (PP Population) | |
| 14.x.2.1.37 | Yes | VWF antigen [%]:Absolute values by subject (PP Population) | |
| 14.x.2.1.38 | Yes | VWF antigen [%]: Absolute values by cohort (PP Population) | |
| 14.x.2.1.39 | Yes | VWF propeptide [mIU/mL]: Absolute values by subject (PP Population) | |
| 14.x.2.1.40 | Yes | VWF propeptide [mIU/mL]: Absolute values by cohort (PP Population) | |
| 14.x.2.1.41 | Yes | Factor VIIIc activity [%]:Absolute values by subject (PP Population) | |
| 14.x.2.1.42 | Yes | Factor VIIIc activity [%]:Absolute values by cohort (PP Population) | |
| 14.x.2.1.43 | Yes | aPTT FS [sec]: Absolute values by subject (PP Population) | |



| 14.x.2.1.44 | Yes | aPTT FS [sec]: Absolute values by cohort (PP | |
|---|---|---|---|
| | | Population) | |
| 14.x.2.1.45 | Yes | Thrombinoscope [nM]: Absolute values by | |
| | | subject (PP Population) | |
| 14.x.2.1.46 | Yes | Thrombinoscope [nM]: Absolute values by | |
| | | cohort (PP Population) | |
| 14.x.2.1.47 | Yes | Fibrin D-dimer [mIU/mL]: Absolute values by | |
| | | subject (PP Population) | |
| 14.x.2.1.48 | Yes | Fibrin D-dimer [mIU/mL]: Absolute values by | |
| | | cohort (PP Population) | |
| 14.x.2.1.49 | Yes | Prothrombin fragment F1.2 [mIU/mL]: | |
| | | Absolute values by subject (PP Population) | |
| 14.x.2.1.50 | Yes | Prothrombin fragment F1.2 [mIU/mL]: | |
| | | Absolute values by cohort (PP Population) | |
| Safety Analys | sis | | |
| 14.x.3.1.40 | Yes | Boxplots of hematology values by group and | Separate figures for every group and |
| | | visit (Safety Population) | every parameter |
| 14.x.3.1.41 | Yes | Boxplots of coagulation values by group and | Separate figures for every group and |
| | | visit (Safety Population) | every parameter |
| 14.x.3.1.42 | Yes | Boxplots of clinical chemistry values by group | Separate figures for every group and |
| | | and visit (Safety Population) | every parameter |
| 14.x.3.1.43 | Yes | Boxplots of urinalysis values by group and | Separate figures for every group and |
| | | visit (Safety Population) | every parameter |
| 14.x.3.1.44 | Yes | Vital signs values by group and visit (Safety | Separate figures for every group and |
| | | Population) | every parameter |
| 14.x.3.1.45 | Yes | ECG values by group and Visit (Safety | Separate figures for every group and |
| | | Population) | every parameter |

# 8. SHELLS OF TABLES, DATA LISTINGS AND FIGURES

For this analysis, no table shells or mock tables are produced, but analysis drafts of TLFs will be generated based on dummy group allocation (dummy randomization list) and dummy immunogenicity data. These drafts will reviewed by the sponsor.